CLINICAL TRIAL: NCT06835335
Title: Differential Opioid Prescribing in the Emergency Department for Patients With Sickle Cell Disease: a Vignette-based International Randomised Trial.
Brief Title: Opioid Prescribing in the Emergency Department for Sickle Cell Disease
Acronym: DOPED-SCD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 25.02.01
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Discrimination, Racial; Pain Management; Emergency Medicine; Sickle Cell Disease
MeSH Terms: conditions — Racism; Agnosia; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-black man: the case will present a non black man
  Interventions: Behavioral: opioid prescription
- Black man: the case will present a non black man
  Interventions: Behavioral: opioid prescription
- non-black woman: the case will present a non black woman
  Interventions: Behavioral: opioid prescription
- black woman: the case will present a black woman
  Interventions: Behavioral: opioid prescription

INTERVENTIONS:
Behavioral: opioid prescription — The intervention consisted of a randomized questionnaire presenting a clinical case of a patient suffering from severe abdominal pain. The control case was "As an emergency physician in an adult emergency department, you are presented with the following patient: The patient is a 39-year-old non-smoking male/female with a history of Meniere's disease and an allergy to Bactrim. He/she presents with abdominal pain that began abruptly 2 hours ago and has persisted despite taking NEFOPAM 45 minutes ago. This is his first episode. His/her vital signs are blood pressure 140/66, heart rate 91, pulse ox 97%, temperature 36.8°C. He/she rates his/her pain as 8/10 without any analgesic position. On clinical examination he/she presents with localized epigastric tenderness. The rest of the abdomen is soft, painless and depressed. There are hydro-aeriform noises. No diarrhea or vomiting. The rest of the clinical examination showed no abnormalities.". In the intervention case, patient had history of S

SUMMARY:
This study consists of a clinical vignette presented to emergency physicians asking them what they would prescribe to a patient with acute abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Being a emergency physician

Exclusion Criteria:

* Working outside of Europe.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population will consist in emergency medicine resident and physician, speaking French or English, in European countries.
  The population will be recruited with the use of professional networks and social medias
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Morphine prescription | through study completion, an average of 1 year
  The proportion of patient for which physician would have prescribed morphine

SECONDARY OUTCOMES:
Analgesic prescription between groups | through study completion, an average of 1 year
  To compare analgesic prescription between groups
factors associated with differences in management between groups | through study completion, an average of 1 year
  identify factors associated with differences in management (urgency level, morphine prescription and computed tomography scan ordering)
Differences according to patient and practitioner gender | through study completion, an average of 1 year
  analyze the difference in morphine treatment prescribed according to patient and practitioner gender

CONTACTS AND LOCATIONS:
Locations (2):
- CHU de Nîmes, Nîmes, Occitanie, France
- Manchester University NHS FT, Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coisy F, Simon A, Occelli C, Dupriez F, Ageron FX, N'Diaye L, Feral-Pierssens AL, Yates G, Bobbia X. Does a history of sickle cell disease affect the prescription of morphine? An international, randomised study based on clinical vignettes conducted among emergency physicians. BMJ Open. 2025 Dec 24;15(12):e108836. doi: 10.1136/bmjopen-2025-108836. PMID 41448706